CLINICAL TRIAL: NCT05133479
Title: Translating Research Into School-based Practice Via Small-group, Language-focused Comprehension Intervention
Brief Title: Let's Know!2: Language-focused Intervention for Children at Risk of Comprehension Difficulties
Acronym: LK!2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MGH Institute of Health Professions (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Ohio State University (Other); University of Kansas (Other)
Responsible Party: Principal Investigator, Tiffany P. Hogan, PhD, CCC-SLP, FASHA, Professor, MGH Institute of Health Professions
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020P002508; 1R01DC018823-01 (NIH)
Record Dates: First submitted 2021-09-10; First posted 2021-11-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Language Disorders in Children
Keywords: language skills; reading comprehension; intervention; specific language impairment; dyslexia
MeSH Terms: conditions — Specific Language Disorder; Dyslexia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive the Let's Know! intervention in small groups as provided by research staff
  Interventions: Behavioral: Let's Know! small-group or TierL 2 Intervention
- Business-As-Usual (No Intervention): Participants continue to receive only their typical classroom instruction (i.e., no small groups)

INTERVENTIONS:
Behavioral: Let's Know! small-group or TierL 2 Intervention — Let's Know!2 is an 22-week intervention spanning 1 school year. Each week features 4, 20-30 minute lessons targeting lower-level and higher-level language skills. Within units, instructors and children progress through specific types of lessons to meet language-focused learning objectives. LK!2 was adapted from the original Let's Know! curriculum (LARRC, 2016). The adaption from LK! to LK! made lessons appropriate for small groups of Grade 1 students with low language skills. Adaptations focused on (1) simplification of language input, (2) increased scaffolding, (3) attention to distributed practice, (4) materials to support diversity and inclusion, and (5) enhanced interventionist training. LK!2 comprised 76 20-30 min lessons across four units (fiction, animals, earth materials, folktales) as implemented by trained research staff (i.e., interventionists).
  Other Names: Let's Know! small-group or Tier 2 Intervention
  Arms: Intervention

SUMMARY:
In the proposed project, the investigators will conduct a multisite randomized controlled trial (RCT) to determine the efficacy of Let's Know!2, a small-group, language focused comprehension intervention, on children's lower- and higher-level language skills and comprehension skills in the short- and long-term (Specific Aims 1 and 2). The investigators will also explore whether intervention effects are moderated by dosage, initial language skill, developmental language disorder (DLD) status, word reading skill, nonverbal IQ, and family socioeconomic status (Specific Aim 3).

Children who have low language skills and are thus at risk for reading comprehension difficulties will participate in the study. Children will be randomly assigned to receive Let's Know! in small groups at their respective schools or to a business-as-usual control condition. The investigators will measure children's language and comprehension skills at the beginning and end of Grade 1 as well as in Grade 2 and Grade 3. The investigators hypothesize that children who experience Let's Know! will end Grade 1 with higher language skills than children in the control condition and that this will translate into better listening and reading comprehension skills as these children matriculate through elementary school.

DETAILED DESCRIPTION:
Parents of children enrolled in Grade 1 at partnering schools will receive consent materials and those who provide consent will complete a brief background/demographic survey about their child. For children whose parents provide informed consent, research staff will (a) ask their educator to confirm basic English proficiency and lack of profound disabilities or behavior issues that severely impair classroom functioning, (b) seek the child's assent to project activities, and (c) administer a language screener in a quiet location at their respective school, either in a small group of other consented children or one-on-one. In order to qualify as eligible for the intervention phase of the study, consented children must: (1) be enrolled in Grade 1 (per educator or parent report) (2) score at or below the empirically derived cut-score on the OWL screener (obtained via direct testing), (3) exhibit at least basic skills in speaking and understanding English (per educator report), (4) not exhibit behavioral difficulties sufficiently severe to prevent participation in the intervention (per educator report), (5) not have a severe disability that would prevent participation in the intervention (per educator report), (6) assent to study activities. Children who meet all eligibility criteria, including scoring below our cutoff on the language screener, will be categorized as potentially eligible for enrollment in the intervention phase of the study. In order to enroll children within a particular school, the investigators must identify a minimum of 6 eligible participants in that school. The investigators will cap the child participants per school at a maximum of 20 in cohort 1 and 10 in cohorts 2 & 3 to allow for later analysis of nested data (children nested within schools; the investigators need 40 schools for appropriate statistical power). Children who are identified as potentially eligible but who attend schools with fewer than 6 total eligible participants, or who consent to the study but have not yet been screened by the time the investigators identify 20 eligible participants in cohort 1 and 10 in cohorts 2 & 3 will be excluded from further participation. In schools in which the investigators have more than the allotted potentially eligible children, the investigators will randomly select the cohort-specific number to enroll in the intervention phase of the study. Children enrolled in the intervention phase of the study will be randomly assigned to receive the Let's Know! intervention or to a business-as-usual control condition. Random assignment will be conducted by Dr. Flemming at KUMC, who will be uninvolved in recruitment, screening, and pretest activities. Prior to intervention start, all enrolled children will complete pretest assessments to measure the lower-level and higher-level language skills targeted by the Let's Know! intervention, comprehension skills, and other abilities (i.e., covariates and moderators for addressing Aim 3). All direct child assessments are listed in Table 1 above. All child direct assessments (screening, pretest, curriculum-aligned measures, posttest, follow-up) will be administered by trained research staff in quiet locations at children's respective schools; alternative arrangements to conduct assessments in the PIs' research laboratories or community locations (e.g., public library) will be made as necessary (e.g., if a child moves into a new, non-partnering school). All but the language screener and Gates-MacGinitie Tests of Reading will be administered individually, with the two exceptions administered to small groups or 1:1, dependent on scheduling. Screening and assessment sessions may be audio or video recorded to allow for accurate scoring and analysis. Following pretest assessments and assignment to conditions, research staff will provide the Let's Know! intervention to small groups of 3 to 5 children allocated to the intervention condition at their respective schools. The Let's Know! intervention provides instruction in the domains of text structure, integration, word knowledge, and grammar; as such, it targets key lower-level (vocabulary) and higher-level (e.g., story grammar, comprehension monitoring, inferencing) language skills to support listening and reading comprehension. The intervention features manualized, soft-scripted lessons that will be provided in small groups of 3-5 children 4 times a week for 25-30 minutes. The lessons are organized into four instructional units that are delivered over 22 weeks. All four instructional units emphasize repeated readings and explorations of commercial texts, with two units comprising narrative books and two comprising expository books. All intervention lessons will be videotaped for purposes of monitoring implementation and coding fidelity. If an individual child misses a session, this will be documented and the session will not be made up. If an entire group misses a session (e.g., due to a field trip/school assembly), the interventionist will wait and deliver that lesson during the next scheduled session (e.g., one group may miss Animals 12 due to a Tuesday assembly; the interventionist teaches Animals 12 at the regularly scheduled Wednesday session and proceeds from there). Children in the control condition will participate in study assessments as noted above but will not experience the Let's Know! intervention. They will receive business-as-usual classroom instruction and supports within their schools. That is, the child's family and school will provide instruction and support for children in the control condition as they typically would for any child not enrolled in the study. The investigators will document the interventions received by children in both the intervention and control conditions.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent to participate in the research;
* Enrollment in Grade 1;
* Scores below the 30th percentile on the OWL Language Screener
* Basic English proficiency as reported by parents/teachers

Exclusion Criteria:

* Unable to speak or understand English at a basic level, as reported by parents/teachers;
* Profound disability that severely impairs classroom participation, as reported by teachers;
* Serious behavior issue that severely impairs classroom participation, as reported by teachers.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment unit 1 (fiction) vocabulary knowledge as assessed by the LARRC Unit Vocabulary Curriculum-Aligned Measure (CAM) total correct | approximately 6 weeks after start of intervention, at the end of Unit 1 treatment
  The Language and Reading Research Consortium (LARRC) Unit Vocabulary Curriculum-Aligned Measure (CAM) assesses children's definitional knowledge of the 8 vocabulary words taught in unit 1 (fiction) and results in a total score of definitional specificity with 2 points possible for each word for a total of 16 points possible.
Treatment unit 2 (animals) vocabulary knowledge as assessed by the LARRC Unit Vocabulary Curriculum-Aligned Measure (CAM) total correct | approximately 12 weeks after start of intervention, at the end of Unit 2 treatment
  The Language and Reading Research Consortium (LARRC) Unit Vocabulary Curriculum-Aligned Measure (CAM) assesses children's definitional knowledge of the 8 vocabulary words taught in unit 2 and results in a total score of definitional specificity with 2 points possible for each word for a total of 16 points possible.
Treatment unit 3 (earth materials) vocabulary knowledge as assessed by the LARRC Unit Vocabulary Curriculum-Aligned Measure (CAM) total correct | approximately 18 weeks after start of intervention, at the end of Unit 3 treatment
  The Language and Reading Research Consortium (LARRC) Unit Vocabulary Curriculum-Aligned Measure (CAM) assesses children's definitional knowledge of the 8 vocabulary words taught in unit 3 and results in a total score of definitional specificity with 2 points possible for each word for a total of 16 points possible.
Treatment unit 4 (folktales) vocabulary knowledge as assessed by the LARRC Unit Vocabulary Curriculum-Aligned Measure (CAM) total correct | approximately 22 weeks after start of intervention, at the end of Unit 4 treatment
  The Language and Reading Research Consortium (LARRC) Unit Vocabulary Curriculum-Aligned Measure (CAM) assesses change in children's definitional knowledge of the 8 vocabulary words taught in unit 4 and results in a total score of definitional specificity with 2 points possible for each word for a total of 16 points possible per CAM.
Change in vocabulary knowledge as assessed by the LARRC Target Word Knowledge | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in vocabulary knowledge as assessed by the Language and Reading Research Consortium (LARRC) Target Word Knowledge measures which assesses definitional knowledge of a sampling of words taught across the 4 treatment units, in addition to several words not taught in the intervention.
Change in breadth of vocabulary as assessed by the Peabody Picture Vocabulary Test 5th Edition (PPVT-5) | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in the breadth of vocabulary will be assessed by the Peabody Picture Vocabulary Test 5th Edition (PPVT-5), a standardized measure of the number of words that a child should know compared to a nationwide sample of age-matched peers. Children point to one picture out of four that best represents a word spoken by the examiner.
Treatment unit 1 (fiction) comprehension monitoring as assessed by the LARRC Unit 1 Comprehension Monitoring Curriculum-Aligned Measure (CAM) | approximately 6 weeks after start of intervention, at the end of Unit 1 treatment
  The Language and Reading Research Consortium (LARRC) Unit 1 (fiction) Comprehension Monitoring Curriculum-Aligned Measure (CAM) assesses children's ability to detect inconsistencies in stories read to them and to recall a strategy to fix their comprehension breakdown.
Treatment unit 2 (animals) comprehension monitoring as assessed by the LARRC Unit 2 Comprehension Monitoring Curriculum-Aligned Measure (CAM) | approximately 12 weeks after start of intervention, at the end of Unit 2 treatment
  The Language and Reading Research Consortium (LARRC) Unit 2 (animals) Comprehension Monitoring Curriculum-Aligned Measure (CAM) assesses children's ability to detect inconsistencies in stories read to them and to recall a strategy to fix their comprehension breakdown.
Treatment unit 3 (earth materials) comprehension monitoring as assessed by the LARRC Unit 3 Comprehension Monitoring Curriculum-Aligned Measure (CAM) | approximately 18 weeks after start of intervention, at the end of Unit 3 treatment
  The Language and Reading Research Consortium (LARRC) Unit 3 (earth materials) Comprehension Monitoring Curriculum-Aligned Measure (CAM) assesses children's ability to detect inconsistencies in stories read to them and to recall a strategy to fix their comprehension breakdown.
Treatment unit 4 (folktales) comprehension monitoring as assessed by the LARRC Unit 4 Comprehension Monitoring Curriculum-Aligned Measure (CAM) | approximately 22 weeks after start of intervention, at the end of Unit 4 treatment
  The Language and Reading Research Consortium (LARRC) Unit 4 (folktales) Comprehension Monitoring Curriculum-Aligned Measure (CAM) assesses children's ability to detect inconsistencies in stories read to them and to recall a strategy to fix their comprehension breakdown.
Change in child's ability to monitoring comprehension, as assessed by the LARRC Comprehension Monitoring Test | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in comprehension monitoring as assessed by the Language and Reading Research Consortium (LARRC) Comprehension Monitoring Test, which assesses child's ability to detect inconsistencies in stories read to them and to recall a strategy to fix their comprehension breakdown from the strategies learned across all 4 treatment units.
Treatment unit 1 (fiction) knowledge of text structures as assessed by the LARRC Unit 1 Text Structure Curriculum-Aligned Measure (CAM) | approximately 6 weeks after start of intervention, at the end of Unit 1 treatment
  The Language and Reading Research Consortium (LARRC) Unit 1 Text Structure Curriculum-Aligned Measure (CAM) assesses children's ability to listen to a story and answer questions about the stories' structure, such as characters, settings, problem, and resolution.
Treatment unit 2 (animals) knowledge of text structures as assessed by the LARRC Unit 2 Text Structure Curriculum-Aligned Measure (CAM) | approximately 12 weeks after start of intervention, at the end of Unit 2 treatment
  The Language and Reading Research Consortium (LARRC) Unit 2 Text Structure Curriculum-Aligned Measure (CAM) assesses children's ability to listen to an expository text passage and answer questions about the passage, such as main idea and important details.
Treatment unit 3 (earth materials) knowledge of text structures as assessed by the LARRC Unit 3 Text Structure Curriculum-Aligned Measure (CAM) | approximately 18 weeks after start of intervention, at the end of Unit 3 treatment
  The Language and Reading Research Consortium (LARRC) Unit 3 Text Structure Curriculum-Aligned Measure (CAM) assesses children's ability to listen to an expository text passage and answer questions about the passage, such as main idea and important details.
Treatment unit 4 (folktales) knowledge of text structures as assessed by the LARRC Unit 1 Text Structure Curriculum-Aligned Measure (CAM) | approximately 22 weeks after start of intervention, at the end of Unit 4 treatment
  The Language and Reading Research Consortium (LARRC) Unit 4 Text Structure Curriculum-Aligned Measure (CAM) assesses children's ability to listen to a story and answer questions about the stories' structure, such as characters, settings, problem, and resolution.
Change in child's ability to use their knowledge to fill in the gaps in short stories, as assessed by the LARRC Inference Task | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in child's ability to use their knowledge to fill in the gaps in short stories, as assessed by the Language and Reading Research Consortium (LARRC) Inference Task, which assesses child's ability to answer questions about short stories they have heard presented by the examiner.
Change in story retelling abilities, as assessed by the CUBED Narrative Retell measure | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in child's ability to accurately and completely retell a story as assessed by the CUBED Narrative Retell measure. The examiner tells the child a story using pictures and the child retells the story back to the examiner.
Change in ability to understand stories, as assessed by the Test of Narrative Language | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in the child's ability to understand stories, as assessed by the Test of Narrative Language. The examiner tells the child stories and asks the child questions about those stories.
Change in a child's ability to comprehend short passages read aloud to them, as assessed by the LARRC Listening Comprehension Measure | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in a child's ability to comprehend short passages read aloud to them, as assessed by the LARRC Listening Comprehension Measure, which requires a child to listen to two short stories and answer questions about those stories
Change in a child's ability to comprehend short passages they read, as assessed by the LARRC Reading Comprehension Measure | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in a child's ability to comprehend short passages they read, as assessed by the LARRC Listening Comprehension Measure, which requires a child to read two short stories and answer questions about those stories
Change in reading comprehension, as assessed by the norm-referenced Gates-McGinitie Reading Test | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in child's ability to comprehend short passages that the child reads to themselves, as assessed by their ability to answer questions about those passages using the norm-referenced Gates-McGinitie Reading Test

OTHER OUTCOMES:
Nonverbal intelligence as assessed by the Kaufman Brief Intelligence Test - Second Edition nonverbal intelligence (matrices) subtest | right before intervention starts
  The nonverbal intelligence (matrices) subtest of the Kaufman Brief Intelligence Test - Second Edition measures children's ability to to solve new problems, perceive relationships and complete visual analogies without taxing language skills. The matrices subtest requires the child to point to the picture that would complete a picture or abstract design. Nonverbal intelligence will be tested as a moderator of treatment effects in analyses.
Change in timed word and nonword reading, as assessed by the Test of Word Reading Efficiency - Second Edition | right before intervention starts, right after intervention ends, one year post intervention, and 2 years post intervention
  Change in timed word and nonword reading accuracy will be assessed by asking children to read as many words and then nonwords as possible in 45 seconds each, as measured by the Test of Word Reading Efficiency - Second Edition. Timed word and nonword reading will be tested as a moderator of treatment effects in the analyses as well as a distal treatment outcome.
Language comprehension skills, as assessed by the OWL Language Screener | right before intervention starts
  Language comprehension skills are assessed by the The OWL Language Screener, which requires children to point to the one picture out of four pictures that best represents a sentence.This measure will be tested as a moderator of treatment effects in analyses as well as the measure to determine if the child has language weaknesses to qualify for treatment.
Academic performance will be assessed by the Massachusetts or Ohio State Assessments of Reading | 2 years after intervention ends
  Children's academic reading performance will be assessed by the Massachusetts or Ohio State Reading Assessments to examine distal treatment outcomes on state assessments of reading

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany P Hogan, PhD, Principal Investigator — MGH Institute of Health Professions
Locations (2):
- United States (2):
  - MGH Institute of Health Professions, Boston, Massachusetts
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goodman WG, Baylink DJ, Sherrard DJ. 24,25(OH)2D3, bone formation, and bone resorption in vitamin D-deficient, azotemic rats. Calcif Tissue Int. 1984 Mar;36(2):206-13. doi: 10.1007/BF02405319. PMID 6430503
- [Background] Adlof, S. M., Catts, H. W., & Little, T. D. (2006). Should the simple view of reading include a fluency component? Reading and Writing: An Interdisciplinary Journal, 19, 933-958.
- [Background] Alloway, T. P., & Gathercole, S. E. (2005). The role of sentence recall in reading and language skills of children with learning difficulties. Learning and Individual Differences, 15, 271-282. doi: https://doi.org/10.1016/j.lindif.2005.05.001
- [Background] Alonzo, C. N., Yeomans-Maldonado, G., Murphy, K. A., Bevens, B., & Language and Reading Research Consortium. (2016). Predicting second grade listening comprehension using prekindergarten measures. Topics in Language Disorders, 36, 312-333.
- [Background] Baumann, J. F., Seifert-Kessell, N., & Jones, L. A. (1992). Effect of think-aloud instruction on elementary students' comprehension monitoring abilities. Journal of Reading Behavior, 24, 143-172.
- [Background] Bengtson, E., Bridges, M., Daniels, D., Brandel, J., & Fisher, C. (2015). Improving language and listening skills in pre-kindergarten children during a summer literacy program. Poster session presented at KSHA, October.
- [Background] Bridges, M.S., Piasta, S., Daniels, D., & Brandel, J. (February, 2016). Small-group intervention to support language and comprehension: Feasibility and Pilot Data. Presented at Pacific Coast Research Conference, San Diego, CA.
- [Background] Castles A, Rastle K, Nation K. Ending the Reading Wars: Reading Acquisition From Novice to Expert. Psychol Sci Public Interest. 2018 Jun;19(1):5-51. doi: 10.1177/1529100618772271. PMID 29890888
- [Background] Catts HW, Nielsen DC, Bridges MS, Liu YS. Early Identification of Reading Comprehension Difficulties. J Learn Disabil. 2016 Sep;49(5):451-65. doi: 10.1177/0022219414556121. Epub 2014 Oct 24. PMID 25344060
- [Background] Catts HW, Adlof SM, Ellis Weismer S. Language deficits in poor comprehenders: a case for the simple view of reading. J Speech Lang Hear Res. 2006 Apr;49(2):278-93. doi: 10.1044/1092-4388(2006/023). PMID 16671844
- [Background] Chall, J. S. (1967). Learning to read: The great debate. New York: McGraw-Hill.
- [Background] Chall, J. S., & Jacobs, V. A. (2003). Poor children's fourth-grade slump. American Educator, 27, 14-15.
- [Background] Ciullo S, Lo YL, Wanzek J, Reed DK. A Synthesis of Research on Informational Text Reading Interventions for Elementary Students With Learning Disabilities. J Learn Disabil. 2016 May-Jun;49(3):257-71. doi: 10.1177/0022219414539566. Epub 2014 Jun 23. PMID 24958632
- [Background] Clements, D. H. (2007). Curriculum research: Toward a framework for research-based curricula. Journal for Research in Mathematics Education, 35-70.
- [Background] Connor CM, Morrison FJ. Individualizing Student Instruction in Reading: Implications for Policy and Practice. Policy Insights Behav Brain Sci. 2016 Mar;3(1):54-61. doi: 10.1177/2372732215624931. Epub 2016 Jan 20. PMID 29732399
- [Background] Coyne, M. D., McCoach, D. B., Loftus, S., Zipoli Jr, R., Ruby, M., Crevecoeur, Y. C., & Kapp, S. (2010). Direct and extended vocabulary instruction in kindergarten: Investigating transfer effects. Journal of Research on Educational Effectiveness, 3, 93-120.
- [Background] Deniz F, Nunez-Elizalde AO, Huth AG, Gallant JL. The Representation of Semantic Information Across Human Cerebral Cortex During Listening Versus Reading Is Invariant to Stimulus Modality. J Neurosci. 2019 Sep 25;39(39):7722-7736. doi: 10.1523/JNEUROSCI.0675-19.2019. Epub 2019 Aug 19. PMID 31427396
- [Background] Dickinson, D. K., Golinkoff, R. M., & Hirsh-Pasek, K. (2010). Speaking out for language:Why language is central to reading development. Educational Researcher, 39, 305-310.
- [Background] Douglas, K., & Albro, E. (2014). The progress and promise of the reading for understanding research initiative. Educational Psychology Review, 26, 341-355.
- [Background] Durlak JA, DuPre EP. Implementation matters: a review of research on the influence of implementation on program outcomes and the factors affecting implementation. Am J Community Psychol. 2008 Jun;41(3-4):327-50. doi: 10.1007/s10464-008-9165-0. PMID 18322790
- [Background] Faggella-Luby, M. N., Drew, S. V., & Schumaker, J. B. (2015). Not such a simple story: Contradictory evidence from a review of story structure research for students at-risk. Learning Disabilities Research & Practice, 30, 61-75.
- [Background] Fien H, Smith JL, Smolkowski K, Baker SK, Nelson NJ, Chaparro E. An Examination of the Efficacy of a Multitiered Intervention on Early Reading Outcomes for First Grade Students at Risk for Reading Difficulties. J Learn Disabil. 2015 Nov-Dec;48(6):602-21. doi: 10.1177/0022219414521664. Epub 2014 Feb 14. PMID 24532827
- [Background] Fixsen, D., Naoom, S., Blase, K., Friedman, R., & Wallace, F. (2005). Implementation research: A synthesis of the literature. Tampa, FL: University of South Florida, Louis de la Parte Florida Mental Health Institute, National Implementation Research Network.
- [Background] Foorman, B., Beyler, N., Borradaile, K., Coyne, M., Denton, C. A., Dimino, J., ... & Keating, B. (2016). Foundational Skills to Support Reading for Understanding in Kindergarten through 3rd Grade. Educator's Practice Guide. NCEE 2016-4008. National Center for Education Evaluation and Regional Assistance.
- [Background] Gates, A. I., & MacGinitie, W. H. (2000). Gates-MacGinitie reading tests (4th ed.). Boston, MA: Riverside.
- [Background] Gersten, R., Fuchs, L. S., Compton, D., Coyne, M., Greenwood, C., & Innocenti, M. S. (2005). Quality indicators for group experimental and quasi-experimental research in special education. Exceptional Children, 71(2), 149-164.
- [Background] Gottfredson DC, Cook TD, Gardner FE, Gorman-Smith D, Howe GW, Sandler IN, Zafft KM. Standards of Evidence for Efficacy, Effectiveness, and Scale-up Research in Prevention Science: Next Generation. Prev Sci. 2015 Oct;16(7):893-926. doi: 10.1007/s11121-015-0555-x. PMID 25846268
- [Background] Hall MS, Burns MK. Meta-analysis of targeted small-group reading interventions. J Sch Psychol. 2018 Feb;66:54-66. doi: 10.1016/j.jsp.2017.11.002. Epub 2017 Nov 15. PMID 29429496
- [Background] Harn BA, Linan-Thompson S, Roberts G. Intensifying instruction: Does additional instructional time make a difference for the most at-risk first graders? J Learn Disabil. 2008 Mar-Apr;41(2):115-25. doi: 10.1177/0022219407313586. PMID 18354932
- [Background] Hebert, M., Bohaty, J. J., Nelson, J. R., & Lambert, M. C. (2018). Identifying and discriminating expository text structures: An experiment with 4th and 5th grade struggling readers. Reading and Writing, 31, 2115-2145.
- [Background] Hogan, T. P., Bridges, M. S., Justice, L. M., & Cain, K. (2011). Increasing higher level language skills to improve reading comprehension. Focus on Exceptional Children, 44, 1-19.
- [Background] Hogan TP, Adlof SM, Alonzo CN. On the importance of listening comprehension. Int J Speech Lang Pathol. 2014 Jun;16(3):199-207. doi: 10.3109/17549507.2014.904441. PMID 24833426
- [Background] Hulme C, Snowling MJ. Learning to Read: What We Know and What We Need to Understand Better. Child Dev Perspect. 2015 Mar 1;7(1):1-5. doi: 10.1111/cdep.12005. PMID 26290678
- [Background] Institute of Education Sciences. (2017, October). What Works Clearinghouse standards handbook (version 4.0). Retrieved August 17, 2018 https://ies.ed.gov/ncee/wwc/Docs/referenceresources/wwc_standards_handbook_v4.pdf
- [Background] Institute of Education Sciences & National Science Foundation. (2013). Common guidelines for education research and development. Washington, DC: Authors.
- [Background] Joseph, L. M., Alber-Morgan, S., Cullen, J., & Rouse, C. (2016). The effects of self-questioning on reading comprehension: A literature review. Reading & Writing Quarterly, 32, 152-173.
- [Background] Kaufman, A. S., & Kaufman, N. L. (1997). Kaufman brief intelligence test (2nd ed.). Minneapolis, MN: NCS Pearson.
- [Background] Language and Reading Research Consortium. (2015). Learning to read: Should we keep things simple? Reading Research Quarterly, 50, 151-169.
- [Background] Language and Reading Research Consortium. (2016). Use of the curriculum research framework (CRF) for developing a reading-comprehension curricular supplement for the primary grades. The Elementary School Journal, 116, 459-486.
- [Background] Language and Reading Research Consortium (LARRC). Oral Language and Listening Comprehension: Same or Different Constructs? J Speech Lang Hear Res. 2017 May 24;60(5):1273-1284. doi: 10.1044/2017_JSLHR-L-16-0039. PMID 28475679
- [Background] Language and Reading Research Consortium, & Chiu, Y. D. (2018). The simple view of reading across development: Prediction of grade 3 reading comprehension from prekindergarten skills. Remedial and Special Education, 39, 289-303. d
- [Background] Language and Reading Research Consortium (LAARC); Farquharson K, Murphy KA. Ten Steps to Conducting a Large, Multi-Site, Longitudinal Investigation of Language and Reading in Young Children. Front Psychol. 2016 Mar 30;7:419. doi: 10.3389/fpsyg.2016.00419. eCollection 2016. PMID 27064308
- [Background] Language and Reading Research Consortium, Jiang, H., & Davis, D. (2017). Let's Know! Proximal impacts on prekindergarten through grade 3 students' comprehension-related skills. The Elementary School Journal, 118, 177-206.
- [Background] Language and Reading Research Consortium (LARRC); Jiang H, Logan JA, Jia R. Modeling the Nature of Grammar and Vocabulary Trajectories From Prekindergarten to Third Grade. J Speech Lang Hear Res. 2018 Apr 17;61(4):910-923. doi: 10.1044/2018_JSLHR-L-17-0090. PMID 29642241
- [Background] Jiang H, Logan J. Improving Reading Comprehension in the Primary Grades: Mediated Effects of a Language-Focused Classroom Intervention. J Speech Lang Hear Res. 2019 Aug 15;62(8):2812-2828. doi: 10.1044/2019_JSLHR-L-19-0015. Epub 2019 Aug 7. PMID 31390289
- [Background] Leslie, L., & Caldwell, J. S. (2011). Qualitative reading inventory (5th ed.). Boston, MA: Pearson.
- [Background] Lohr, S., Schochet, P.Z., & Sanders, E (2014). Partially Nested Randomized Controlled Trials in Education Research: A Guide to Design and Analysis. (NCER 2014-2000). Washington, DC: U.S. Department of Education, Institute of Education Sciences, National Center for Educational Research.
- [Background] Lonigan, C. J., Burgess, S. R., & Schatschneider, C. (2018). Examining the simple view of reading with elementary school children: Still simple after all these years. Remedial and Special Education, 39, 260-273.
- [Background] McNeish D, Stapleton LM. Modeling Clustered Data with Very Few Clusters. Multivariate Behav Res. 2016 Jul-Aug;51(4):495-518. doi: 10.1080/00273171.2016.1167008. Epub 2016 Jun 7. PMID 27269278
- [Background] Moir, T. (2018). Why is implementation science important for intervention design and evaluation within educational settings? Frontiers in Education, 3.
- [Background] Morris ZS, Wooding S, Grant J. The answer is 17 years, what is the question: understanding time lags in translational research. J R Soc Med. 2011 Dec;104(12):510-20. doi: 10.1258/jrsm.2011.110180. PMID 22179294
- [Background] Nation, K. (2001). Reading and language in children: Exposing hidden deficits. The Psychologist, 14(5), 238-242.
- [Background] Nation K, Adams JW, Bowyer-Crane CA, Snowling MJ. Working memory deficits in poor comprehenders reflect underlying language impairments. J Exp Child Psychol. 1999 Jun;73(2):139-58. doi: 10.1006/jecp.1999.2498. PMID 10328862
- [Background] Nation K, Clarke P, Marshall CM, Durand M. Hidden language impairments in children: parallels between poor reading comprehension and specific language impairment? J Speech Lang Hear Res. 2004 Feb;47(1):199-211. doi: 10.1044/1092-4388(2004/017). PMID 15072539
- [Background] Norbury CF, Gooch D, Wray C, Baird G, Charman T, Simonoff E, Vamvakas G, Pickles A. The impact of nonverbal ability on prevalence and clinical presentation of language disorder: evidence from a population study. J Child Psychol Psychiatry. 2016 Nov;57(11):1247-1257. doi: 10.1111/jcpp.12573. Epub 2016 May 16. PMID 27184709
- [Background] Pearson, P. D., & Gallagher, M. C. (1983). The instruction of reading comprehension. Contemporary educational psychology, 8(3), 317-344.
- [Background] Petscher Y, Justice LM, Hogan T. Modeling the Early Language Trajectory of Language Development When the Measures Change and Its Relation to Poor Reading Comprehension. Child Dev. 2018 Nov;89(6):2136-2156. doi: 10.1111/cdev.12880. Epub 2017 Jul 5. PMID 28677872
- [Background] Phillips BM, Tabulda G, Ingrole SA, Burris PW, Sedgwick TK, Chen S. Literate Language Intervention With High-Need Prekindergarten Children: A Randomized Trial. J Speech Lang Hear Res. 2016 Dec 1;59(6):1409-1420. doi: 10.1044/2016_JSLHR-L-15-0155. PMID 27960007
- [Background] Phillips BM, Zhao Y, Weekley MJ. Teacher language in the preschool classroom: Initial validation of a classroom environment observation tool. Early Educ Dev. 2018;29(3):379-397. doi: 10.1080/10409289.2017.1408371. Epub 2017 Dec 13. PMID 32189955
- [Background] Piasta, S. B., Farley, K. S., Mauck, S. A., Soto Ramirez, P., Schachter, R. E., O'Connell, A. A., . . . Weber-Mayrer, M. (in press). At-scale, state-sponsored language and literacy professional development: Impacts on early childhood classroom practices and children's outcomes. Journal of Educational Psychology.
- [Background] Piasta, S. B., Logan, J. A. R., Groom, L. J., Zettler-Greeley, C. M., Bailet, L. L., & Lewis, K. (2019). Implementation of a small-group emergent literacy intervention by preschool teachers and community aides. Manuscript submitted for publication.
- [Background] Quinn, D. M., & Kim, J. S. (2017). Scaffolding fidelity and adaptation in educational program implementation: Experimental evidence from a literacy intervention. American Educational Research Journal, 54, 1187-1220.
- [Background] ead-e Set Grow. (2013). Predictive assessment of reading: Pre-k to grade 3 edition. Clemmons, NC: Author.
- [Background] Redmond SM, Ash AC, Christopulos TT, Pfaff T. Diagnostic Accuracy of Sentence Recall and Past Tense Measures for Identifying Children's Language Impairments. J Speech Lang Hear Res. 2019 Jul 15;62(7):2438-2454. doi: 10.1044/2019_JSLHR-L-18-0388. Epub 2019 Jun 20. PMID 31220421
- [Background] Ritchie SJ, Bates TC. Enduring links from childhood mathematics and reading achievement to adult socioeconomic status. Psychol Sci. 2013 Jul 1;24(7):1301-8. doi: 10.1177/0956797612466268. Epub 2013 May 2. PMID 23640065
- [Background] Rudd, A., & Johnson, R. B. (2008). Lessons learned from the use of randomized and quasiexperimental field designs for the evaluation of educational programs. Studies in Educational Evaluation, 34, 180-188.
- [Background] Sanetti, L. M. H. T. R. (2009). Toward developing a science of treatment integrity: Introduction to the special series. School Psychology Review, 38, 445.
- [Background] Semel, E., Wiig, E. H., & Secord, W. A. (2003). Clinical evaluation of language fundamentals:4. San Antonio, TX: The Psychological Corporation.
- [Background] Shadish, W. R., Cook, T. D., & Campbell, D. T. (2002). Experimental and quasi-experimental designs for generalized causal inference. New York: Houghton Mifflin.
- [Background] Silverman, R., & Crandell, J. D. (2010). Vocabulary practices in prekindergarten and kindergarten classrooms. Reading Research Quarterly, 45(3), 318-340.
- [Background] Torgesen, J. K. (2000). Individual differences in response to early interventions in reading: The lingering problem of treatment resisters. Learning Disabilities Research & Practice, 15(1), 55-64.
- [Background] Torgesen, J. K., Wagner, R. K., & Rashotte, C. A. (1999). Test of word reading efficiency. Austin, TX: Pro-Ed.
- [Background] Vaughn, S., Linan-Thompson, S., Kouzekanani, K., Pedrotty Bryant, D., Dickson, S., & Blozis, S.A. (2003). Reading instruction grouping for students with reading difficulties. Remedial and Special Education, 24, 301-315.
- [Background] Wright, T. S., & Cervetti, G. N. (2017). A systematic review of the research on vocabulary instruction that impacts text comprehension. Reading Research Quarterly, 52, 203-226
- [Background] Wright, T. S., & Neuman, S. B. (2013). Vocabulary instruction in commonly used kindergarten core reading curricula. The Elementary School Journal, 113(3), 386-408.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT05133479/Prot_ICF_000.pdf